CLINICAL TRIAL: NCT06458569
Title: Employment of Natural Killer Opioid Receptor as a Biomarker to Ameliorate the Efficacy of the Rehabilitation Program in a Patient-oriented Strategy
Brief Title: NK-ORB Expression of Mu Receptor on Lymphocytes in Rehabilitation
Acronym: NK-ORB
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 22/30
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia
Keywords: Chronic Pain, NK cells, Lymphocytes, Mu Opioid Receptor
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples from patients in EDTA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy subjects: subjects with NRS<5
- patients with cronical pain: patients with NRS>5
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — 3-weeks rehabilitation in hospital
  Groups: patients with cronical pain

SUMMARY:
Chronic pain is a serious disorder that causes physical suffering and emotional distress.

NK cells are cytotoxic granular cells playing a crucial role in innate immunity.

Recent studies described modulation of the percentage of B lymphocytes and NK cells expressing the μ opioid receptor as a potential marker for measuring pain. Neuropathic pain sufferers have decreased NK cell function, highlighting the need of further investigating the effect of opioid receptor expression on lympoid cells defining their potential relevance as a pain monitor marker. Opioid receptors expressed on NK, B and T cells are a possible candidate for objective monitoring of pain in patients.

DETAILED DESCRIPTION:
Pain is a serious global problem Based on the preliminary data, peripheral blood of pain suffering patients who have entered a neurorehabilitation program will be investigated to confirm the modulation of the percentage of Mu-positive NK cells and to evaluate if they could be eligible as predictive markers of chronic pain.

All patients in the experimental group will undergo three blood sample collections at specific time points to evaluate the percentage of Mu-positive NK cells, and its modulation according to rehabilitation programs: the day of the enrollment (T0), at half part of the neuro rehabilitation programs (T1) and at the end of neuro-rehabilitation programs (T2). Particularly, the two study groups involved will be in a experimental group (50 consecutive patients who have an NRS >5); a control group (50 patients who have an NRS <5).

Peripheral blood will be incubated with different fluorochrome-conjugated antibodies, specific for natural killer cells, in combination with anti-Mu Opioid Receptor (MOR) and the data will be analyze usin flow cytometer and FlowJo. The level of statistical significance will be fixed at p < 0.05. Analyses will be carried out using GraphPad Prism software (v8.00; GraphPad Software). The results are expressed as mean ± SEM The expected results from this study could support the hypothesis that modulation of the µ opioid receptor on NK cells is a valid method for pain measurement, helping to establish an innovative approach in a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

IRCCS San Raffaele Roma patients who entered the neuro-rehabilitation program, aged 18 years older, able to sign a written informed consent.

Exclusion Criteria:

* Patients with oncological or psychiatric diseases.
* Pregnant patients
* Patients with a severe psychiatric disorder (excluding mild depression) or mental/cognitive impairment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Experimental group, patients who have an NRS >5;
  * Control group, patients who have an NRS <5.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Identification of percentage of Mu-positive NK cells as predictive markers of pain in suffering patients | 3 weeks
  Peripheral blood of pain suffering patients who have entered a neurorehabilitation program will be investigated to confirm the modulation of the percentage of Mu-positive NK cells and to evaluate if they could be eligible as predictive markers of chronic pain by correlating it to the level of pain calculated with Numeric Pain Rating Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Roma, Italy